CLINICAL TRIAL: NCT04654871
Title: Effects of Glucosamine and Chondroitin Sulfate Supplementation in Addition to Resistance Exercise Training and Manual Therapy in Patients With Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FUI/CTR/2020/11
Record Dates: First submitted 2020-11-26; First posted 2020-12-04 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-12

CONDITIONS: Osteoarthritis; Osteoarthritis, Knee
Keywords: chondroitin sulfate; resistance exercise; strength training; manual therapy; glucosamine; joint mobilization
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Knee | interventions — Chondroitin Sulfates; Resistance Training; Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental)
  Interventions: Dietary Supplement: Chondroitin Sulfate; Procedure: Resistance exercise training; Procedure: Manual therapy / Joint Mobilization; Procedure: THE therapy
- Active Comparator Group (Experimental)
  Interventions: Procedure: Resistance exercise training; Procedure: Manual therapy / Joint Mobilization; Procedure: THE therapy

INTERVENTIONS:
Dietary Supplement: Chondroitin Sulfate — Glucosamine 500 mg Chondroitin sulfate sodium 400mg 3/day
  Arms: Experimental Group
Procedure: Resistance exercise training — Treadmill walking 5-10 min for warm up Strength training: (80% of 8RM)
  Supervised exercise thrice a week and Home Exercise 4 times a week Leg press knee extension Knee flexion Terminal knee extension Mini squats 3 sets 8 reps 10-15 s rep rest interval 1-2 min set rest interval
Procedure: Manual therapy / Joint Mobilization — Ant. tib-fem glide Post tib-fem glide thrice a week Pattelo-femoral joint mobilization
Procedure: THE therapy — Interferential and Heating for 20 min

SUMMARY:
Osteoarthritis (OA) IS one of the most common joint disorders, affecting not only the joints but also the surrounding muscles, which become weak. Resistance exercise reduces pain and improves function in patients with OA of the knee. Nonsteroidal anti-inflammatory drugs (NSAIDs) are widely used by patients with OA to reduce pain and thereby maintain the ability to perform daily activities. However, there is accumulating evidence for a negative effect of NSAIDs, thus many patients with OA are treated with dietary supplementations such as glucosamine and chondroitin sulfate, and some studies show a beneficial effects on cartilage and pain. However, their effect on OA symptoms and cartilage remains controversial. Thus, it is important to investigate whether a potentially beneficial effect of glucosamine and chondroitin sulfate with resistance exercise and manual therapy in patients with knee OA.

ELIGIBILITY:
Inclusion Criteria:

* knee osteoarthritis for at least 3 months
* knee pain no more than 8/10
* Grade III or less on radiograph (Kellgren classification)

Exclusion Criteria:

* Malignancy
* Any additional Inflammatory disorders
* Infection
* Knee trauma
* lower limb fracture
* Lumbar radiculopathy or myelopathy
* knee surgery or replacement
* Intra-articular steroid therapy in the last 2 months

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | 2 weeks
  Visual Analogue Scale was used to measure pain scoring from 0-10 cm on a horizontal 10cm line. A greater score reflects higher pain intensity.
Visual Analogue Scale | 4 weeks
  Visual Analogue Scale was used to measure pain scoring from 0-10 cm on a horizontal 10cm line. A greater score reflects higher pain intensity.
Knee Injury and Osteoarthritis Outcome Score | 2 weeks
  Knee Injury and Osteoarthritis Outcome Score (KOOS) to measure physical function and quality of life. A greater score on Knee Injury and Osteoarthritis Outcome Score reflects good prognosis and outcome and a lower score shows poor prognosis and outcome. the score for Knee Injury and Osteoarthritis Outcome Score is reported in the form of percentage i.e. 0-100%.
Knee Injury and Osteoarthritis Outcome Score | 4 weeks
  Knee Injury and Osteoarthritis Outcome Score (KOOS) to measure physical function and quality of life. A greater score on Knee Injury and Osteoarthritis Outcome Score reflects good prognosis and outcome and a lower score shows poor prognosis and outcome. the score for Knee Injury and Osteoarthritis Outcome Score is reported in the form of percentage i.e. 0-100%.
Knee Joint Range of Motion | 2 weeks
  Knee Joint Range of Motion will be measured via goniometry. It is a continuous scale and a greater score reflects greater angular movement possible at the knee joint, which is measured in degrees.
Knee Joint Range of Motion | 4 weeks
  Knee Joint Range of Motion will be measured via goniometry. It is a continuous scale and a greater score reflects greater angular movement possible at the knee joint, which is measured in degrees.
Body Composition | 2 weeks
  Body Composition was measured via bioelectrical impedance analysis. A greater Phase angle reflects better cellular integrity and smaller phase angle reflects poorer cellular integrity.
Body Composition | 4 weeks
  Body Composition was measured via bioelectrical impedance analysis. A greater Phase angle reflects better cellular integrity and smaller phase angle reflects poorer cellular integrity.
Fall risk | 2 weeks
  Fall risk will be measured via Biodex balance system, and greater score reflects greater fall risk and poorer outcome.
Fall risk | 4 weeks
  Fall risk will be measured via Biodex balance system, and greater score reflects greater fall risk and poorer outcome.
5 repetition sit to stand test | 2 weeks
  Time will be measured to perform 5 repetitions of sit to stand activity. Lesser time means a better score.
5 repetition sit to stand test | 4 weeks
  Time will be measured to perform 5 repetitions of sit to stand activity. Lesser time means a better score.
Modified sphygmomanometer dynamometry | 2 weeks
  Modified sphygmomanometer dynamometry was used to measure muscle strength. Greater score will reflect greater muscle strength. The unit of Modified sphygmomanometer dynamometry used will be mmHg (millimeter of mercury).
Modified sphygmomanometer dynamometry | 4 weeks
  Modified sphygmomanometer dynamometry was used to measure muscle strength. Greater score will reflect greater muscle strength. The unit of Modified sphygmomanometer dynamometry used will be mmHg (millimeter of mercury).

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University Institute of Rehabilitation Sciences., Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Osama M, Babur MN, Siddiqi FA, Tassadaq N, Arshad Tareen MA. Effects of glucosamine and chondroitin sulfate supplementation in addition to resistance exercise training and manual therapy in patients with knee osteoarthritis: A randomized controlled trial. J Pak Med Assoc. 2022 Jul;72(7):1272-1277. doi: 10.47391/JPMA.2444. PMID 36156542